CLINICAL TRIAL: NCT01100866
Title: Randomized Controlled Trial of POMELLA™ Extract in Prostate Cancer Patients Scheduled for Surgery
Brief Title: Study of POMELLA™ Extract to Treat Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to slow enrollment
Sponsor: Vancouver Coastal Health (Other Government)
Collaborators: Lotte & John Hecht Memorial Foundation (Other)
Responsible Party: Principal Investigator, Dr. Alan I. So, Principal Investigator, Vancouver Coastal Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PML-01054
Record Dates: First submitted 2010-04-02; First posted 2010-04-09 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: clinically localized Prostate Cancer; low and intermediate risk for relapse; candidates for radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): POMELLA™ 2 x 500mg capsule once daily
  Interventions: Dietary Supplement: POMELLA™ (pomegranate extract)
- Group 2 (Placebo Comparator): POMELLA™ placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: POMELLA™ (pomegranate extract) — in a capsule form, 2 x 500mg once daily
  Other Names: POMELLA™
  Arms: Group 1
Other: Placebo — placebo capsules
  Arms: Group 2

SUMMARY:
This is a randomized, two-arm, placebo controlled trial to evaluate benefit of treatment using POMELLA™ extract on mechanisms known to drive prostate cancer. This research allows provision for biochemical and histological comparisons to be made between POMELLA™ treated and placebo treated prostate tissues removed from men with organ confined prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men 18 years or older (19 years in BC) with a histologic diagnosis of clinically localized prostate cancer prior to radical prostatectomy as defined by:

  1. Clinical state T1-T2
  2. PSA <20
  3. Gleason score ≤ 7
* ECOG performance status of 0-1.
* Life expectancy greater than 10 years.
* Able to understand and give informed consent.
* Laboratory values must be as follows:

  1. White blood cell count: ≥ 3,000/mm^3
  2. Absolute granulocyte count: ≥ 1,500/mm^3
  3. Platelets: ≥ 100,000/mm^3
  4. Hemoglobin: ≥ 12g/dL
  5. Serum creatinine: ≤ 1.5 x ULN
  6. AST: ≤ 2 x ULN
  7. ALT: ≤ 2 x ULN
  8. Serum calcium: ≤ ULN
  9. Total bilirubin: ≤ 1.5 x ULN

Exclusion Criteria:

* Patients who are receiving any other investigational therapy.
* Patients who have received or are receiving any other treatment for their prostate cancer.
* Patients with an active serious infection or other serious underlying medical condition that would otherwise impair their ability to receive protocol treatment.
* Dementia or significantly altered mental status that would prohibit the understanding and/or giving of informed consent.
* Histologic evidence of small cell carcinoma of the prostate.
* Patients who are currently receiving active therapy for other neoplastic disorders will not be eligible for study.
* Patients who are receiving any androgens, estrogens or progestational agents.
* Patients with a known hypersensitivity to pomegranates or composites of the capsules/placebo: hydroxypropyl methylcellulose, silicon dioxide or aerosol.
* Patients who are taking any drugs or natural health products which might impact biochemical tests (some examples include: spironolactone, aprepitant, bexarotene, clarithromycin, itraconazole, ketoconazole, St. John's wort). A washout period of 30 days prior to commencing the study would be necessary for these compounds if required.
* Patients who have chronic active hepatitis.
* Medical conditions, which, in the opinion of the investigators would jeopardize either the patient or the integrity of the data obtained.

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Tissue collection and Bioanalysis of the specimens collected | Tissue collected on Day 31 (after 30 days of study treatment)
  Prostate tissue are collected at radical radical prostatectomy. These specimens are used to explore the effects of treatment on the expression of the proliferation markers, enzymes, hormnes, receptors and cell signaling proteins known to influence prostate cancer progression.

CONTACTS AND LOCATIONS:
Overall Officials: Alan I So, MD, FRCSC, Principal Investigator — Vancouver Coastal Health
Locations (1):
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada